CLINICAL TRIAL: NCT06007963
Title: Impella Left or Right Ventricular Support in Cardiogenic Shock
Brief Title: Impella in Cardiogenic Shock Registry
Acronym: Impella
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 62048
Record Dates: First submitted 2019-04-03; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2022-12

CONDITIONS: Shock, Cardiogenic
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Coagulation tests
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment with impella device. — Impella percutaneous mechanical supported patients will be included after revision to support.

SUMMARY:
The purpose of the study is to evaluate the safety, efficacy and clinical usefulness of a mechanical support strategy with the impella device.

DETAILED DESCRIPTION:
In the last two decades mortality from acute coronary syndromes has decreased dramatically thanks to aggressive use of coronary revascularization techniques. In cardiogenic shock however, a dramatique decrease in mortality since the introduction of primary PCI has not been seen, probably because restoring only coronary flow does not necessary imply restoration of whole body organ perfusion as long as the heart has not recuperated. To restore perfusion there are currently two options: catecholamine drugs (that can increase native cardiac output but at the price of increased oxygen consumption by the myocardium) or mechanical cardiac support (which provides artificial blood flow to the body, but depending on the device increases or decreases myocardial oxygen consumption). The dose of catecholamines used in cardiogenic shock patients is linearly correlated with worse outcome, suggesting a negative effect. Several mechanical cardiac support devices have been developed, but only some can be placed percutaneously and are available in Belgium.

The intra-aortic balloon pump, which was the first and remains the least invasive device, failed to show any mortality benefit in cardiogenic shock. A possible explanation could be the fact that this device device aims at restoring coronary rather than organ perfusion, since the increase in cardiac output after starting the balloon pump is very limited. Extracorporeal membrane oxygenation (ECMO) is an alternative to support organ perfusion, that provides the highest blood flow, but tends to increase cardiac work because it increases afterload. ECMO is also the most invasive percutaneous device since this requires two large bore access catheters to the patients' circulation and the blood flows through a bigger circuit, making it more prone to coagulation defects. The left side Impella device is a micro-axial continuous flow pump which sucks blood from the left ventricle towards the ascending aorta with the goal of increasing blood flow to the body while at the same time unloading the heart. This device only requires one access site (mostly smaller caliber as well). There is extensive experience with the left sided Impella device; its safety and efficacy have already been demonstrated in the past. The first results of the recent 'Detroit Cardiogenic Shock Initiative', aiming at early institution of mechanical support with the Impella device, already showed a significant decrease in mortality in participating centers. The Impella RP device is one of the only percutaneous devices that provide high flow support to the right ventricle by pushing blood from the inferior vena cava to the pulmonary artery. In the FDA approval study safety was demonstrated and outcomes where significantly better with the devices compared to historical controls.

An evolution to an earlier and as minimally invasive as possible strategy for mechanical support in cardiogenic shock is seen as well in the UZ Leuven cardiac intensive care unit. With an expierience of more than 20 years with the impella device in UZ Leuven (among the first to use the earlier versions of the device) this device was chosen as the first step to support the heart (in case of failure of one ventricle without need for additional oxygenation), with ECMO in second line since it is more invasive but delivers biventricular support with capability of higher flows. There are no high quality randomized controlled trials that compare one mechanical support strategy to another (except for one study in which almost 90% of patients were included after cardiac arrest, mostly dying from withdrawal of therapy). To improve quality, it seems key to measure outcomes and analyze these results as thoroughly as possible. For this reason, a prospective registry for all cardiogenic shock patients in the cardiac ICU, treated with the Impella device, is started.

ELIGIBILITY:
Inclusion Criteria:

* • Patients admitted for cardiogenic shock (defined as SBP <90 mmHg without vasopressors/inotropics or elevated serum lactate).

AND

• Treatment with Impella device

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A/ Awake patients will only be asked for consent after getting oral and written information.
  B/ Ventilated patients will be included after consent is obtained from legal representative. After improvent of patients status consent will be obtained from the patient.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 day and 1 year
  Description: mortality: as assessed via patient file, contact with patient, general physician or family memeber

SECONDARY OUTCOMES:
Myocardial recovery | 30 dat and 1 year
  myocardial recovery: assesses as the difference between echocardiographic left ventricular ejection fracton assessment (baseline versus follow-up time point)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Adriaenssens, MD PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Gasthuisberg, Leuven, Belgium